CLINICAL TRIAL: NCT01895569
Title: Effects on Glycemic Variability and Glyco-metabolic Control of Metformin, Pioglitazone and Sitagliptin in Type 2 Diabetic Patients
Brief Title: Triple Therapy in Type 2 Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, MD, PhD, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120021548
Record Dates: First submitted 2013-06-30; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Pioglitazone; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Type 2 diabetic patients (Experimental): Type 2 diabetic patients, naive to treatment, and not well controlled by diet (glycate hemoglobin > 6.5%, and < 9.0%) will be instructed to take metformin, followed by metformin plus pioglitazone, and then metformin plus pioglitazone plus sitagliptin.
  Interventions: Drug: Metformin; Drug: Pioglitazone; Drug: Sitagliptin

INTERVENTIONS:
Drug: Metformin — Metformin will be added to therapy for the first threre months.
  Other Names: 500 mg three times a day
Drug: Pioglitazone — In patients not well controlled (glycated hemoglobin >6.5%) after three months of metformin, pioglitazone will be added.
  Other Names: 15 mg twice a day
Drug: Sitagliptin — In patients not well controlled (glycated hemoglobin >6.5%) after three months of metformin and pioglitazone, sitagliptin will be added.
  Other Names: 100 mg once a day

SUMMARY:
The treatment of type 2 diabetes mellitus often requires the use of one or more hypoglycemic agents to reach the adequate glycemic control. The aim of the study is to evaluate the effects of a triple therapy with metformin, pioglitazone and sitagliptin on glycemic variability compared to metformin monotherapy, and compared to a combination of metformin and pioglitazone. To assess glycemic variability a continuous glucose monitoring system will be used.

DETAILED DESCRIPTION:
In an estimated temporal space of about 3 years, 64 not well controlled, type 2 diabetic patients will be recruited.

Patients will be instructed to take metformin 500 mg three times a day for the first three months, then pioglitazone 15 mg twice a day will be added for further three months, and finally sitagliptin 100 mg once a day will be added for the last three months. At the baseline, and every three months a continuous glucose monitoring system will be performed.

At any stage of the study, if the value of glycated hemoglobin reach the desired goal (<6.5%), participation in the study will be stopped and the patient will not be subjected to further adjustments of hypoglycemic therapy or additional continuous monitoring glucose.

After collection of written informed consent, the following data will be collected:

* History: type of diabetes, comorbidities, current medication, duration of diabetes and complications, voluptuary habits such as tobacco smoke (both number of packets/year and n° packets/day), alcohol consumption, coffee consumption, physical activity.
* Physical exam, general anthropometric parameters such as weight, height, circumference, body mass index, waist-hip ratio, and blood pressure.
* Assessment of glycemic variability every three months using a continuous glucose monitoring system.
* Collection of blood and urine samples to assess: glycated hemoglobin, fasting plasma glucose (FPG), post-prandial glucose (PPG), fasting plasma insulin (FPI), HOMA-index (HOMA-IR and HOMA-β), high sensitivity C-reactive protein (hs-CRP), total cholesterol, LDL-cholesterol, HDL-cholesterol, tryglicerides, lipoprotein (a) [Lp(a)], metalloproteinase-2 (MMP-2), metalloproteinase-9 (MMP-9), soluble adhesion molecules (sICAM-1, sVCAM-1), sE-selectin, adiponectin (ADN), complete urinalysis, 24-hour microalbuminuria.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients
* naive to therapy
* glycated hemoglobin > 6.5 and < 9.0 %

Exclusion Criteria:

* hepatic and renal diseases
* recent cardiovascular diseases
* previous pancreatitis
* history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Glycemic variability | 9 months
  Glycemic variability will be assessed at the baseline, and every three months, using a continuous glucose monitoring system.

SECONDARY OUTCOMES:
Glyco-metabolic control | 9 months
  Glyco-metabolic control will be assessed evaluating glycated hemoglobin, fasting plasma glucose and post-prandial glucose.

OTHER OUTCOMES:
Insulin-resistance parameters | 9 months
  Insulin-resistance parameters will be assessed using HOMA-index (HOMA-IR and HOMA-β).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, PhD, Principal Investigator — IRCCS Policlinico San Matteo Foundation
Locations (1):
- IRCCS Policlinico S. Matteo Foundation, Pavia, Italy